CLINICAL TRIAL: NCT06813911
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Pelacarsen (TQJ230) With Background Inclisiran in Participants With Atherosclerotic Cardiovascular Disease (ASCVD), and Elevated LDL-C and Lp(a)
Brief Title: Lp(a) Lowering Study of Pelacarsen (TQJ230) With Background Inclisiran in Participants With Elevated Lp(a) and Established ASCVD
Acronym: ADD-VANTAGE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTQJ230A12304
Expanded Access: NCT07000695 (Available)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Atherosclerotic Cardiovascular Disease (ASCVD)
Keywords: Lipoprotein(a); cardiovascular disease; ASCVD; pelacarsen (TQJ230)
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases | interventions — pelacarsen; ALN-PCS

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pelacarsen (Active Comparator): Participants randomized in Pelacarsen arm, will be administered pelacarsen (TQJ230) subcutaneous injection once monthly for 12 months.
  Interventions: Drug: Pelacarsen; Drug: Inclisiran
- Placebo (Placebo Comparator): Participants will be administered placebo subcutaneous injection once monthly for 6 months. After Month 6, all participants will receive pelacarsen 80 mg injection for the remaining 6 months during the open-label treatment period.
  Interventions: Drug: Pelacarsen; Drug: Placebo; Drug: Inclisiran

INTERVENTIONS:
Drug: Pelacarsen — Pelacarsen will be provided as solution for injection in prefilled syringe 80 mg for subcutaneous injection.
  Other Names: TQJ230
Drug: Placebo — Placebo will be provided as solution for injection in prefilled syringe for subcutaneous injection.
  Arms: Placebo
Drug: Inclisiran — All participants will be administered two loading doses of inclisiran as background treatment at Run-in 1 and Run-in 2, separated by 3 months, according to the approved label. After that inclisiran will be administered every 6 months, i.e., Month 5 and Month 11.

SUMMARY:
The purpose of the study CTQJ230A12304, is to evaluate the efficacy, safety, and tolerability of pelacarsen (TQJ230) compared to placebo in participants with ASCVD who have elevated lipoprotein(a) (Lp(a)), and who are on background inclisiran treatment for elevated low-density lipoprotein cholesterol (LDL-C).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter, parallel group study followed by an open-label treatment period.

ELIGIBILITY:
Key Inclusion criteria:

* Male and female participants 18 to ≤80 years of age at Screening visit
* Established ASCVD, defined as documented coronary heart disease (CHD), cerebrovascular disease (CVD), or peripheral arterial disease (PAD) at Screening visit
* On stable dose of local guideline recommended lipid lowering therapy for at least 30 days prior to Screening visit
* Participants must successfully complete the run-in period of background inclisiran treatment in order to be randomized
* On standard of care (SoC) treatment for other CVD risk factors including hypertension and diabetes for at least 30 days prior to Randomization/Baseline visit
* Central laboratory reported Lp(a) ≥175 nmol/L at Screening visit
* Central laboratory reported LDL-C >70 mg/dL (or >1.8 mmol/L) at Screening visit

Key Exclusion Criteria:

* Prior treatment with inclisiran
* Any other PCSK9 inhibitor (e.g., evolocumab, alirocumab) use within 4 months prior to Screening visit
* Uncontrolled hypertension at Randomization/Baseline visit
* Heart failure New York Heart Association (NYHA) class IV at Screening visit or at Randomization/Baseline visit (Day 1)
* Triglycerides ≥400 mg/dL at Screening visit
* History of malignancy of any organ system within the past 5 years
* Myocardial infarction, stroke or other major bleeding, coronary or lower limb re vascularization, major cardiac or non-cardiac surgery between Screening visit and Randomization/Baseline visit (Day 1)
* Central laboratory reported platelet count <140,000 per mm3
* Active liver disease or hepatic dysfunction at Screening visit
* Significant kidney disease at Screening visit
* Pregnant or nursing women at Screening visit
* Any uncontrolled chronic or serious medical condition which may pose an immediate risk to clinical stability of the study participant at Screening visit

  * Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-11-05 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in log transformed lipoprotein A (Lp(a)) concentration | Baseline, 6 Months
  To evaluate the efficacy of Pelacarsen compared to placebo, in reducing Lp(a) levels at Month 6 in ASCVD participants who have elevated Lp(a), and who are on background inclisiran for elevated LDL-C

SECONDARY OUTCOMES:
Proportion of participants achieving reduction in Lp(a) levels at Month 6 | Baseline, Month 6
  Efficacy of pelacarsen versus placebo in reducing Lp(a)
Incidence of treatment emergent adverse events (TEAEs) and treatment emergent serious adverse events (TESAEs) | 16 Months
  The TEAEs will be defined as any recorded AE with start date located in the on-treatment period. To understand the effect of pelacarsen versus placebo on safety and tolerability in participants treated with background inclisiran. Incidence and severity of AEs by treatment group, including changes in the vital signs, electrocardiogram and laboratory results qualifying and reported as AEs.
Incidence of treatment emergent adverse events of special interest (AESI) | 12 Months
  To understand the effect of pelacarsen versus placebo on safety and tolerability in participants treated with background inclisiran
Incidence of study and treatment discontinuations due to TEAEs | 12 Months
  Incidence proportion of study discontinuations due to TEAEs

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (48):
- United States (32):
  - Parkway Medical Center, Birmingham, Alabama
  - Clinical Research Inst of Arizona, Sun City West, Arizona
  - National Heart Institute, Beverly Hills, California
  - Interv Cardiology Med Grp, West Hills, California
  - Excel Medical Clinical Trials LLC, Boca Raton, Florida
  - Jacksonville Center for Clinical, Jacksonville, Florida
  - University of Miami Hospital, Miami, Florida
  - Miami Cancer Institute at Bapt, Miami, Florida
  - Inpatient Research Clinical LLC, Miami Lakes, Florida
  - FXM Clin Res Miramar LLC, Miramar, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - SEC Clinical Research, Pensacola, Florida
  - Peace River Cardiovascular Center, Port Charlotte, Florida
  - FC Site Partners Miami, Winter Park, Florida
  - Advocate Lutheran General Childrens Hospital, Park Ridge, Illinois
  - American Health Network Research Dept, Muncie, Indiana
  - Cardiovascular Associates Research, Covington, Louisiana
  - Omega Clinical Research, Metairie, Louisiana
  - Anderson Medical Research, Ft. Washington, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Aa Mrc Llc, Flint, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - AB Clinical Trials, Las Vegas, Nevada
  - Overlook Medical Center, Summit, New Jersey
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - The Corvallis Clinic P C, Corvallis, Oregon
  - Novartis Investigative Site, Tullahoma, Tennessee
  - PharmaTex Research LLC, Amarillo, Texas
  - Kelsey Seybold Research Foundation, Houston, Texas
  - Northwest Houston Clinical Research PLLC, Tomball, Texas
  - Intermountain Medical Center, Murray, Utah
  - Virginia Heart, Falls Church, Virginia
- China (5):
  - Novartis Investigative Site, Yinchuan, Ningxia
  - Novartis Investigative Site, Jining, Shandong
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- Hong Kong (2):
  - Novartis Investigative Site, Hong Kong, Hong Kong
  - Novartis Investigative Site, Hong Kong
- Latin Clinical Trial Center Inc, San Juan, Puerto Rico
- Taiwan (4):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- United Kingdom (4):
  - Novartis Investigative Site, Chichester, West Sussex
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Tyne and Wear

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Novartis.aspx